CLINICAL TRIAL: NCT02547597
Title: Comparison of Carvedilol and Atenolol on Anti-anginal and Metabolic Effects in Patients With Stable Angina Pectoris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Woong Chol Kang, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARVEDILOL
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-09

CONDITIONS: Stable Angina Pectoris
Keywords: Beta-blockers; Anti-anginal effect; Lipid metabolism; Glucose metabolism
MeSH Terms: conditions — Angina, Stable | interventions — Carvedilol; Atenolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol 25 mg twice a day
  Interventions: Drug: Carvedilol
- Atenolol (Active Comparator): Atenolol 50 mg twice a day
  Interventions: Drug: Atenolol

INTERVENTIONS:
Drug: Carvedilol
  Arms: Carvedilol
Drug: Atenolol
  Arms: Atenolol

SUMMARY:
There are few data regarding anti-anginal effects between beta-blockers with and without vasodilating property. Beta-blocker without vasodilating property is generally known to have unfavorable effects on glucose and lipid metabolism. Therefore, the investigators compared carvedilol and atenolol on anti-anginal and metabolic effects in patient with stable angina pectoris.

DETAILED DESCRIPTION:
Previous studies have demonstrated that beta-blockers are effective in reducing not only ischemia but also cardiovascular mortality following myocardial infarction. And, recent guidelines have suggested the potential for use of beta-blockers as first-line agents in chronic stable angina. However, beta-blockers are a diverse class with different mechanisms of action and physiological effects. Various pharmacologic properties that characterize beta-blockers include cardioselectivity, intrinsic sympathomimetic activity, and concomitant vasodilating alpha-adrenoceptor blockade, which might exhibit differential anti-anginal efficacies. In addition, traditional beta-blockers, particularly nonvasodilating beta-blockers, have been reported to have negative metabolic effects, including hyperglycemia, insulin resistance, and dyslipidemia. These unfavorable effects of beta-blockers should be considered in patients with stable angina pectoris, because the pathophysiology of coronary artery disease is associated with abnormalities in glucose and lipid metabolism. Carvedilol, a newer vasodilating beta-blocker, has been shown to differ from traditional beta-blockers in terms of metabolic effects in patients with hypertension and diabetes. However, few data regarding comparative anti-anginal and metabolic effects between beta-blockers with and without vasodilating property have been reported, particularly in patients with angina pectoris. In this study, we simultaneously compared anti-anginal and metabolic effects of carvedilol and atenolol in patients with stable angina pectoris.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina pectoris who had a positive exercise treadmill test according to the American College of Cardiology Foundation and the American Heart Association guidelines

Exclusion Criteria:

* Acute coronary syndrome
* Coronary revascularization within the past 3 months
* Asthma or chronic obstructive lung disease
* Bradycardia (heart rate < 55 beat/min)
* History of severe adverse reaction to beta-blockers
* Symptomatic arrhythmia requiring anti-arrhythmia therapy
* Heart failure
* Severe renal or hepatic failure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Time to 1-mm ST-segment depression | After 25 weeks of treatment
  Time to 1-mm ST-segment depression at exercise treadmill test
Time to onset of angina | After 25 weeks of treatment
  Time to onset of angina at exercise treadmill test

SECONDARY OUTCOMES:
Blood pressure at resting and peak exercise | After 25 weeks of treatment
  Blood pressure at resting and peak exercise during exercise treadmill test
Heart rate at resting and peak exercise | After 25 weeks of treatment
  Heart rate at resting and peak exercise during exercise treadmill test
Lipid profiles | After 25 weeks of treatment
  Lipid profiles: total cholesterol, triglyceride, high-density lipoprotein-cholesterol, and low-density lipoprotein-cholesterol
Glucose metabolism | After 25 weeks of treatment
  Fasting glucose, insulin, HbA1c, Quantitative Insulin-Sensitivity Check Index (QUICKI)
Seattle Angina Questionnaire (SAQ) scores | After 25 weeks of treatment
Treatment-emergent adverse events | After 25 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

REFERENCES:
- [Derived] Oh PC, Kang WC, Moon J, Park YM, Kim S, Kim MG, Lee K, Ahn T, Shin EK. Anti-Anginal and Metabolic Effects of Carvedilol and Atenolol in Patients with Stable Angina Pectoris: A Prospective, Randomized, Parallel, Open-Label Study. Am J Cardiovasc Drugs. 2016 Jun;16(3):221-8. doi: 10.1007/s40256-016-0168-1. PMID 27021556